CLINICAL TRIAL: NCT04306315
Title: Adjustable Brodalumab Dosage Regimen Compared With Standard Brodalumab Treatment for 52 Weeks in Subjects With Moderate-to-severe Plaque Psoriasis and ≥120 kg Body Weight
Brief Title: Adjusted Brodalumab Dose Compared With Standard Brodalumab Dose in Subjects With Moderate-to-severe Plaque Psoriasis and ≥120 kg Body Weight
Acronym: ADJUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0160-1329; 2017-004998-13 (EudraCT Number); U1111-1282-4507 (Other: World Health Organization (WHO)); 2023-509668-11-00 (EU CTIS Number)
Record Dates: First submitted 2020-03-11; First posted 2020-03-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pre-filled syringes with 210 mg (1.5 mL) brodalumab will be open-label. The packaging and labelling of the pre-filled syringes with 70 mg (0.5 mL) brodalumab or placebo will contain no evidence to distinguish brodalumab from placebo. It is not considered possible to distinguish between brodalumab and placebo visually; both solutions are colourless.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Brodalumab 210 mg + brodalumab 70 mg add-on* (adjusted brodalumab dosing regimen) (Experimental): Participants will receive 210 mg brodalumab subcutaneously at Week 0, Week 1, and Week 2, and then once every 2 weeks. *Participants not fulfilling a predefined response at any visit with efficacy assessments after Week 16 will receive a dose adjustment to 280 mg brodalumab every 2 weeks.
  Interventions: Biological: Brodalumab
- Brodalumab 210 mg + placebo add-on* (standard brodalumab treatment) (Placebo Comparator): Participants will receive 210 mg brodalumab subcutaneously at Week 0, Week 1, and Week 2, and then once every 2 weeks. *Participants not fulfilling a predefined response at any time visit with efficacy assessments Week 16 will receive a dose adjustment to 210 mg brodalumab + placebo every 2 weeks.
  Interventions: Biological: Brodalumab

INTERVENTIONS:
Biological: Brodalumab — Brodalumab is an anti-IL-17 receptor antibody, which blocks the inflammatory effects of IL-17 in the skin.

SUMMARY:
This study investigates if an adjusted brodalumab dosage regimen will give improved efficacy in psoriasis in patients with a body weight of over 120 kg. The increased dosage regimen will be compared to the standard brodalumab treatment plus placebo.

DETAILED DESCRIPTION:
Brodalumab is an anti-IL-17 receptor antibody and blocks the inflammatory effects of IL-17 in the skin. Some psoriasis patients with a higher body weight experienced a lower treatment effect of brodalumab in clinical studies. Therefore, the purpose of this study is to investigate if increasing the dose of brodalumab will increase the effect of treatment for patients with a higher body weight. The study will run over 60-62 weeks, including screening, treatment period and safety follow-up, with the primary endpoint measurement at Week 40. Patients will receive subcutaneous injections of brodalumab at Week 0, 1, and 2, followed by injections every 2 weeks. Participants not fulfilling a predefined response at any time after Week 16 will receive a dose adjustment to 280 mg brodalumab or 210 mg brodalumab plus placebo every 2 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed and dated informed consent has been obtained prior to any protocol-related procedures.
* Age ≥18 to <75 years at the time of screening.
* Diagnosed with chronic plaque psoriasis at least 6 months before randomisation.
* Body weight ≥120 kg at the time of screening.
* Moderate-to-severe plaque psoriasis as defined by: BSA ≥10% and PASI ≥12 at screening and baseline.
* No evidence of active or latent tuberculosis according to local standard of care.

Key Exclusion Criteria:

* Diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, or other skin conditions (e.g., eczema) that would interfere with evaluations of the effect of the investigational medicinal product (IMP) on participants with plaque psoriasis.
* Clinically important active infections or infestations, chronic, recurrent or latent infections or infestations, or is immunocompromised (e.g., human immunodeficiency virus, hepatitis B, and hepatitis C).
* Any systemic disease considered by the investigator to be uncontrolled and either immunocompromising the participants and/or placing the participant at undue risk of intercurrent diseases (including, but not limited to, renal failure, heart failure, liver disease, diabetes, and anaemia).
* History of Crohn's disease.
* Myocardial infarction or stroke, or unstable angina pectoris within the past 12 months.
* Any active malignancy.
* History of malignancy within 5 years, except for treated and considered cured cutaneous squamous or basal cell carcinoma, in situ cervical cancer, or in situ breast ductal carcinoma.
* History of suicidal behaviour (i.e., 'actual suicide attempt', 'interrupted attempt', 'aborted attempt', or 'preparatory acts or behaviour') based on the Columbia-Suicide Severity Rating Scale (C-SSRS) questionnaire at screening or at baseline.
* Any suicidal ideation of category 4 or 5 ('active suicidal ideation with some intent to act, without specific plan' or ' active suicidal ideation with specific plan and intent') based on the C-SSRS questionnaire at screening or at baseline.
* A Patient Health Questionnaire (PHQ)-8 score of ≥10 corresponding to moderate-to-severe depression at screening or at baseline.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Having at least 90% lower Psoriasis Area and Severity Index (PASI) score relative to baseline (PASI 90 response) at Week 40. | Week 40
  The PASI score is the most widely used tool in clinical practice and clinical trials to assess the severity and extent of psoriasis. The assessment is done based on the condition of the disease at the time of evaluation and not in relation to the condition at a previous visit. The investigator will assess the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions, head/neck, trunk, upper extremities, and lower extremities, according to a severity scale. The investigator will also assess the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0-72, with higher values indicating a more severe and/or more extensive condition.

SECONDARY OUTCOMES:
Having static Physician's Global Assessment (sPGA) score of 0 or 1 at Week 40 | Week 40
  The sPGA is an instrument used in clinical trials to rate the severity of the participant's global psoriasis and is based on a 6-point scale ranging from 0 (clear) to 5 (very severe).
Having PASI 90 response at Week 52 | Week 52
  The PASI score is the most widely used tool in clinical practice and clinical trials to assess the severity and extent of psoriasis. The assessment is done based on the condition of the disease at the time of evaluation and not in relation to the condition at a previous visit. The investigator will assess the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions, head/neck, trunk, upper extremities, and lower extremities, according to a severity scale. The investigator will also assess the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0-72, with higher values indicating a more severe and/or more extensive condition. PASI 90 is defined as at least 90% improvement in PASI relative to baseline.
Having sPGA score of 0 or 1 at Week 52 | Week 52
  The sPGA is an instrument used in clinical trials to rate the severity of the participant's global psoriasis and is based on a 6-point scale ranging from 0 (clear) to 5 (very severe).
Having sPGA of genitalia (sPGA-G) score of 0 or 1 at both Week 40 and Week 52 | Week 40
  The sPGA-G score is based on a combination of erythema and the secondary features (plaque elevation and/or scale) and it is used to rate the severity of the participant's psoriasis of the genitalia on a 6-point scale ranging from 0 (clear) to 5 (very severe).
Having sPGA of genitalia (sPGA-G) score of 0 or 1 at Week 40 | Week 40
  The sPGA-G score is based on a combination of erythema and the secondary features (plaque elevation and/or scale) and it is used to rate the severity of the participant's psoriasis of the genitalia on a 6-point scale ranging from 0 (clear) to 5 (very severe).
Having sPGA-G score of 0 or 1 at Week 52 | Week 52
  The sPGA-G score is based on a combination of erythema and the secondary features (plaque elevation and/or scale) and it is used to rate the severity of the participant's psoriasis of the genitalia on a 6-point scale ranging from 0 (clear) to 5 (very severe).
Having PASI 100 response at Week 40 | Week 40
  The PASI score is the most widely used tool in clinical practice and clinical trials to assess the severity and extent of psoriasis. The assessment is done based on the condition of the disease at the time of evaluation and not in relation to the condition at a previous visit. The investigator will assess the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions, head/neck, trunk, upper extremities, and lower extremities, according to a severity scale. The investigator will also assess the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0-72, with higher values indicating a more severe and/or more extensive condition. PASI 100 is defined as 100% improvement in PASI relative to baseline.
Having PASI 100 response at Week 52 | Week 52
  The PASI score is the most widely used tool in clinical practice and clinical trials to assess the severity and extent of psoriasis. The assessment is done based on the condition of the disease at the time of evaluation and not in relation to the condition at a previous visit. The investigator will assess the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions, head/neck, trunk, upper extremities, and lower extremities, according to a severity scale. The investigator will also assess the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0-72, with higher values indicating a more severe and/or more extensive condition. PASI 100 is defined as 100% improvement in PASI relative to baseline.
Change from baseline at Weeks 40 and 52 in PASI score | Week 40 and 52
  The PASI score is the most widely used tool in clinical practice and clinical trials to assess the severity and extent of psoriasis. The assessment is done based on the condition of the disease at the time of evaluation and not in relation to the condition at a previous visit. The investigator will assess the severity of 3 psoriasis disease characteristics (redness, thickness, and scaliness) on each of the 4 body regions, head/neck, trunk, upper extremities, and lower extremities, according to a severity scale. The investigator will also assess the extent of psoriasis within each of the 4 body regions. This gives a composite score ranging from 0-72, with higher values indicating a more severe and/or more extensive condition.
Change from baseline at Weeks 40 and 52 in affected body surface area (BSA) | Week 40 and 52
  To assess the full BSA with psoriatic involvement, the investigator will use the surface area of the participant's hand (palm and fingers) as a reference measurement to determine the percentage of the body surface area that is affected by psoriasis. One hand is approximately equal to 1% total BSA.
Having Dermatology Life Quality Index (DLQI) total score of 0 or 1 at Week 40 | Week 40
  The Dermatology Life Quality Index (DLQI) is a validated questionnaire with content specific to those with dermatology conditions. The DLQI consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their HQoL over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all ⁄not relevant'; 1 = 'a little'; 2 = 'a lot'; 3 = 'very much'). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor HQoL.
Having DLQI total score of 0 or 1 at Week 52 | Week 52
  The Dermatology Life Quality Index (DLQI) is a validated questionnaire with content specific to those with dermatology conditions. The DLQI consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their HQoL over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all ⁄not relevant'; 1 = 'a little'; 2 = 'a lot'; 3 = 'very much'). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor HQoL.
Change from baseline at Weeks 40 and 52 in DLQI total score | Week 40 and 52
  The Dermatology Life Quality Index (DLQI) is a validated questionnaire with content specific to those with dermatology conditions. The DLQI consists of 10 items addressing the participant's perception of the impact of their skin disease on different aspects of their health-related quality of life (HrQoL) over the last week such as dermatology-related symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the treatment (10). Each item is scored on a 4-point Likert scale (0 = 'not at all ⁄not relevant'; 1 = 'a little'; 2 = 'a lot'; 3 = 'very much'). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor HrQoL.
Number of Participants Experiencing Adverse Events (AEs) up to Week 58. | Week 58

CONTACTS AND LOCATIONS:
Overall Officials: Medical Medical Expert, Study Director — LEO Pharma
Locations (68):
- Belgium (4):
  - LEO Pharma Investigational Site, Brussels
  - LEO Pharma Investigational Site, Ham-sur-Heure-Nalinnes
  - LEO Pharma Investigational Site, Leuven
  - LEO Pharma Investigational Site, Liège
- Czechia (3):
  - LEO Pharma Investigational Site, Kutná Hora
  - LEO Pharma Investigational Site, Nový Jičín
  - LEO Pharma Investigational Site, Plzen-Bory
- France (4):
  - LEO Pharma Investigational Site, Amiens, Somme
  - LEO Pharma Investigational Site, Saint-Priest-en-Jarez
  - LEO Pharma Investigational Site, Toulouse
  - LEO Pharma Investigational Site, Valence
- Germany (14):
  - LEO Pharma Investigational Site, Langenau, Baden-Wurttemberg
  - LEO Pharma Investigational Site, Limburg an der Lahn, Hesse
  - LEO Pharma Investigational Site, Wiesbaden, Hesse
  - LEO Pharma Investigational Site, Lohne, Lower Saxony
  - LEO Pharma Investigational Site, Mainz, Rhineland-Palatinate
  - LEO Pharma Investigational Site, Kiel, Schleswig-Holstein
  - LEO Pharma Investigational Site, Berlin, State of Berlin
  - LEO Pharma Investigational Site, Bad Bentheim
  - LEO Pharma Investigational Site, Bielefeld
  - LEO Pharma Investigational Site, Hamburg
  - LEO Pharma Investigational Site, Memmingen
  - LEO Pharma Investigational Site, Münster
  - LEO Pharma Investigational Site, Oldenburg
  - LEO Pharma Investigational Site, Osnabrück
- Greece (4):
  - LEO Pharma Investigational Site, Heraklion, Crete
  - LEO Pharma Investigational Site, Athens
  - LEO Pharma Investigational Site, Piraeus
  - LEO Pharma Investigational Site, Thessaloniki
- Hungary (4):
  - LEO Pharma Investigational Site, Debrecen
  - LEO Pharma Investigational Site, Orosháza
  - LEO Pharma Investigational Site, Szolnok
  - LEO Pharma Investigational Site, Veszprém
- Italy (10):
  - LEO Pharma Investigational Site, Ancona
  - LEO Pharma Investigational Site, Bologna
  - LEO Pharma Investigational Site, Brescia
  - LEO Pharma Investigational Site, Coppito
  - LEO Pharma Investigational Site, Modena
  - LEO Pharma Investigational Site, Napoli
  - LEO Pharma Investigational Site, Parma
  - LEO Pharma Investigational Site, Pavia
  - LEO Pharma Investigational Site, Roma
  - LEO Pharma Investigational Site, Rozzano
- LEO Pharma Investigational Site, Beek, Netherlands
- Poland (7):
  - LEO Pharma Investigational Site, Iwonicz-Zdrój
  - LEO Pharma Investigational Site, Lodz
  - LEO Pharma Investigational Site, Lublin
  - LEO Pharma Investigational Site, Poznan
  - LEO Pharma Investigational Site, Skierniewice
  - LEO Pharma Investigational Site, Warsaw
  - LEO Pharma Investigational Site, Wroclaw
- Spain (10):
  - LEO Pharma Investigational Site, Alicante
  - LEO Pharma Investigational Site, Badalona
  - LEO Pharma Investigational Site, Barcelona
  - LEO Pharma Investigational Site, Granada
  - LEO Pharma Investigational Site, Manises
  - LEO Pharma Investigational Site, Pontevedra
  - LEO Pharma Investigational Site, Pozuelo de Alarcón
  - LEO Pharma Investigational Site, Santiago de Compostela
  - LEO Pharma Investigational Site, Valencia
  - LEO Pharma Investigational Site, Villajoyosa
- United Kingdom (7):
  - LEO Pharma Investigational Site, Chorley
  - LEO Pharma Investigational Site, Corby
  - LEO Pharma Investigational Site, Coventry
  - LEO Pharma Investigational Site, Liverpool
  - LEO Pharma Investigational Site, London
  - LEO Pharma Investigational Site, Northwood
  - LEO Pharma Investigational Site, Shipley

IPD SHARING:
Plan to Share IPD: No